CLINICAL TRIAL: NCT03727906
Title: Sleep and Cardiovascular Health in Adolescence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SRI International (Industry)
Responsible Party: Principal Investigator, Massimiliano de Zambotti, Research Scientist, SRI International
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 50116
Record Dates: First submitted 2018-10-25; First posted 2018-11-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Insomnia Type; Sleep Disorder
Keywords: Cardiovascular; Blood Pressure; ECG; EEG
MeSH Terms: conditions — Sleep Wake Disorders | interventions — BaseLine dental cement

STUDY DESIGN:
Intervention Model Description: The experimental paradigm will consist of three in-lab counterbalanced non-consecutive (≥2 days in-between) polysomnography (PSG) nights in which we will modulate the level of pre-sleep psychophysiological arousal in a group of insomnia and non-insomnia adolescents.
  1. no pre-sleep arousal manipulation night;
  2. pre-sleep arousal down-regulation night (pre-sleep relaxation-driven Virtual reality ANS downregulation);
  3. pre-sleep arousal up-regulation night (pre-sleep anticipation of stress using the Trier Social StressTest).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-insomnia Group (Other): Non-insomnia participants will not meet criteria for current DSM-5 Insomnia Disorder or have a past history of insomnia.
  Interventions (order is randomly assigned):
  1. no pre-sleep arousal manipulation night;
  2. pre-sleep arousal down-regulation night
  3. pre-sleep arousal up-regulation night.
  Interventions: Other: No pre-sleep arousal manipulation; Other: pre-sleep arousal down-regulation; Other: pre-sleep arousal up-regulation
- Insomnia Group (Other): Insomnia Group participants will have to meet DSM-5 criteria for current Insomnia Disorder.
  Interventions (order is randomly assigned):
  1. no pre-sleep arousal manipulation night;
  2. pre-sleep arousal down-regulation night
  3. pre-sleep arousal up-regulation night.
  Interventions: Other: No pre-sleep arousal manipulation; Other: pre-sleep arousal down-regulation; Other: pre-sleep arousal up-regulation

INTERVENTIONS:
Other: No pre-sleep arousal manipulation — As with the pre-sleep arousal up- and down-regulation nights, the participant will sleep in comfortable sound-proof and temperature-controlled bedroom and will go to bed and wake up at his/her self-reported usual school-week times. On this night, pre-sleep activities include watching television or reading a book.
  Other Names: Baseline
Other: pre-sleep arousal down-regulation — On the "low pre-sleep arousal night", about 30 min before lights-out, a 20 min session of relaxation-driven Virtual Reality (VR) + slow breathing will be conducted. Adolescents will be instructed to perform slow diaphragmatic breathing and to let the VR immersion guide them through this relaxation process.
  Other Names: pre-sleep relaxation
Other: pre-sleep arousal up-regulation — On the "high pre-sleep arousal" night, an anticipatory stress procedure from the Trier Social Stress Test (TSST) will be used to elicit stress-induced ANS activation in the pre-sleep period. About 30 min before lights-out participants will be told that the following morning they will need to prepare and give a 5-min speech in front of a panel of assessors who will judge their performance and ask questions. Participants will be shown the testing room (set up with chairs, video camera, microphone).
  Other Names: pre-sleep stress

SUMMARY:
Insomnia is a prevalent and under-recognized disorder in adolescence, particularly in girls, with long-term repercussions for mental and physical health. This study assesses manifestation of autonomic hyperarousal and vulnerability to insomnia using a sample of male and female adolescents with and without Diagnostic and Statistical Manual (DSM-5) Insomnia Disorder. Outcomes from this study have the potential to inform prevention and treatment interventions for insomnia that can be implemented at a young age before chronic negative sequelae of this common disorder manifest.

DETAILED DESCRIPTION:
Insomnia is highly prevalent in adolescence, particularly in post-pubertal girls and tends to persist over time. Insomnia is considered a hyperarousal disorder, in which abnormally elevated levels of cognitive and physiological activation, particularly evident at bed-time, prevent individuals from falling asleep and having a restorative night's sleep. Hyperarousal is a major pathophysiological mechanism linking insomnia with poor mental and physical health, including cardiovascular (CV) disease. The investigators and others have shown evidence of autonomic nervous system (ANS) dysfunction such as hyperactivation of the sympathetic branch of the ANS - a major etiological factor in CV disease - in young and midlife adults, both before and during sleep. It is unknown if ANS hyperarousal is evident in adolescents with insomnia.

The biological basis for an emerging sex difference in insomnia prevalence in adolescence is unknown. The investigators' pilot data reveal intriguing evidence of sex-differences in basic and stress-dependent ANS modulation during sleep in adolescents with girls showing a greater ANS response to stress. These data suggest the existence of a predisposing and stress-dependent ANS vulnerability in female adolescents, a potential pathway to develop insomnia. This study takes a novel approach to investigating the manifestation of physiological ANS and CV hyperarousal in adolescents with insomnia by experimentally manipulating the pre-sleep arousal state via stress-induced ANS up-regulation and relaxation-driven ANS down-regulation. In addition, the study focuses on sex differences in ANS and CV responses to pre-sleep ANS manipulation, potentially addressing the question of why female sex is a major risk factor for insomnia.

The investigators aim to test 110 male and female high-school students (16-20y) with and without DSM-5 Insomnia Disorder, during a regular in-lab polysomnographic night (baseline) and under experimental pre-sleep stress (psychosocial stressor) and pre-sleep relaxation (Virtual reality ANS bio-feedback) intervention nights, using state-of-the-art, noninvasive, beat-to-beat ANS and CV measures, including blood pressure, to assess nocturnal ANS and CV function in adolescents with insomnia (Aim 1); the impact of pre-sleep ANS arousal levels on nocturnal ANS and CV function, and sleep in adolescents with and without insomnia, considering possible sex differences (Aim 2), and the extent to which nocturnal ANS and CV function mediate the effect of pre-sleep arousal levels on objective and perceived sleep quality (Aim 3).

This study has the potential to elucidate pathophysiological ANS hyperarousal underlying Insomnia Disorder in adolescence, including potential reasons for the vulnerability to insomnia in girls, leading to better recognition and potentially new treatment strategies of this disorder targeted at the state of ANS hyperarousal in the pre-sleep period.

ELIGIBILITY:
Inclusion Criteria:

* Must be post-pubertal
* BMI <30 kg/m-2 to reduce the likelihood of obesity-related sleep-disordered breathing

Exclusion Criteria:

* Current use of drugs known to affect sleep and CV systems (e.g., Antidepressants, stimulants, beta-blockers)
* Serious history of, or current medical conditions that could affect brain function, or study participation, including Diabetes, cancer, neurological diseases (e.g., Seizure disorders) recurrent migraine, cardiovascular diseases (e.g., Hypertension) and traumatic brain injury with loss of consciousness >30 minutes
* Current DSM-5 diagnosis of Neurodevelopmental Disorders (e.g., Attention-Deficit/Hyperactivity Disorder)
* Current DSM-5 diagnosis of Schizophrenia Spectrum and Other Psychotic Disorders, Bipolar and Related Disorders
* Current DSM-5 diagnosis of Depressive and Anxiety Disorders (e.g., Major Depressive Disorder)
* Current DSM-5 diagnosis of Post-Traumatic Stress Disorder
* Current DSM-5 diagnosis of Substance-Related and Addictive Disorders (e.g., Alcohol Use Disorder)
* History of and persistence in severe learning disorder, pervasive developmental disorder, or other condition requiring repeated or persistent specialized education (e.g., Estimated intellectual quotient (IQ) >2 standard deviations below mean)
* Current psychiatric disorders in both control and insomnia groups is exclusionary
* Past history of psychiatric disorders in controls is exclusionary (past history of psychiatric disorders in the insomnia group is not exclusionary)
* Shift work in the previous year and no time-zone travel in the past month
* Evidence of other DSM-5 Sleep-Wake Disorders (e.g., Narcolepsy), Breathing-Related Sleep Disorders (e.g., Obstructive Sleep Apnea Hypopnea, Circadian Rhythm Sleep-Wake Disorders and particularly Delayed Sleep Phase Type), and Parasomnias (e.g., Non-Rapid Eye Movement Sleep Arousal Disorders, Rapid Eye Movement Sleep Behavior Disorder and Restless Legs Syndrome)
* Current pregnancy

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 115 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-08-27 (Actual)

PRIMARY OUTCOMES:
Average nocturnal heart rate (HR), as a measure of cardiac contractility | Measured during 1 night (each for baseline, pre-sleep stress and pre-sleep relaxation conditions)
  Heart rate (HR) response to experimental manipulation
Average nocturnal Pre-ejection period (PEP), as a measure of cardiac sympathetic activity | Measured during 1 night (each for baseline, pre-sleep stress and pre-sleep relaxation conditions)
  Pre-ejection period (PEP) response to experimental manipulation

CONTACTS AND LOCATIONS:
Locations (1):
- SRI International, Menlo Park, California, United States